CLINICAL TRIAL: NCT05204992
Title: Effectiveness of Ultrasound Guided Hydro-dissection of Median Nerve in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Ahmed ElSadek (Unknown); Iman Hamed (Unknown)
Responsible Party: Principal Investigator, Mai Fathy Ahmed Fahmy, Lecturer of Neurology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R 154/2021
Record Dates: First submitted 2022-01-07; First posted 2022-01-24 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrodissection (Experimental): ultrasound guided hydrodissection
  Interventions: Procedure: ultrasound guided hydrodissection

INTERVENTIONS:
Procedure: ultrasound guided hydrodissection — Injection of steroids, saline and bupivicaine ultrasound guided

SUMMARY:
60 patients with carpal tunnel syndrome will undergo ultrasound guided hydrodissection of the median nerve with follow up using Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) at 3, 6 and 12 months

DETAILED DESCRIPTION:
Aim of study:

to evaluate the effectiveness of ultrasound guided hydrodissection of median nerve as minimal invasive procedure in carpal tunnel syndrome

Study Design:

60 patients with a clinical diagnosis of mild-to moderate CTS will be evaluated clinically and confirmed by neurophysiological study (NCV and EMG study). patients will undergo ultrasound guided hydrodissection, from the outpatient clinic of Neurology department, Ain shams University hospitals.

Study Subjects:

Our subjects aged 25-65 years with clinical diagnosis of mild to moderate CTS .

Patients will be assessed using Boston Carpal Tunnel Syndrome Questionnaire. Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS, which encompasses 2 components(4). In total, 11 questions and 8 items were evaluated for rating on the Symptom Severity Scale (SSS) and Functional Status Scale (FSS), respectively. Both subscales score from 1 to 5, with a higher score indicating a greater degree of disability.

Subjects will be excluded if they met any of this exclusion criteria: Pregnancy, Cancer, hypothyroidism , systemic infection, history of polyneuropathy, cervical radiculopathy, brachial plexopathy, thoracic outlet syndrome , history of previous carpal tunnel open surgery or local steroid injection and severe CTS (confirmed by el electrophysiological studies)

Ultrasound-guided hydrodissection using ultrasonography (MyLab 5, Esaote, Italy) with a 5-10 MHZ linear array probe will be done by the same experienced doctor. The probe is placed in the flexor surface of the wrist at pisiform-scaphoid level to detect median nerve at the inlet of carpal tunnel with the probe oriented in the transverse (anatomic axial ) plane of carpal tunnel. A 25-guage needle is inserted from ulnar side advancing to the radial side via the in-plane approach. Hydrodissection fluid( 5 cc normal saline, 2 ml steroids, 1 ml bupivicaine) is injected in the plane between median nerve and transverse carpal ligament to separate the nerve from the deep surface of flexor retinaculum (using the jet of injected fluid from the needle tip)

Primary outcome:

Change from baseline of severity of symptoms and functional status on 3rd , 6th and 12 months month after injection [ Time Frame: Pre-treatment, 3rd,6th and 12th month after injection ] using Boston Carpal Tunnel Syndrome Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical diagnosis of mild to moderate CTS and confirmed by neurophysiological studies.
* The clinical symptoms and signs of CTS are as follows:

  1. sensory symptoms in the form of paresthesia, dysesthesia, pain and numbness of the hand in the distribution of median nerve which was more nocturnal, postural or related to hand overuse and relieved by frequent shaking of the hand
  2. motor symptoms in the form of decreased strength of the thenar muscles
  3. positive Phalen and/or Tinel sign.

Exclusion Criteria:

* Pregnancy
* Cancer
* hypothyroidism
* systemic infection
* history of polyneuropathy
* cervical radiculopathy
* brachial plexopathy
* thoracic outlet syndrome
* history of previous carpal tunnel open surgery or local steroid injection and severe CTS (confirmed by el electrophysiological studies)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | 12 months
  Boston Carpal Tunnel Syndrome Questionnaire, highest score is 95, lowest score is 19, higher score denotes worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided